CLINICAL TRIAL: NCT06689709
Title: Determination Of Serum Alkaline Phosphatase Levels In Healthy Turkish Children
Brief Title: Serum Alkaline Phosphatase Levels In Healthy Turkish Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Hafize (Other)
Responsible Party: Sponsor-Investigator, Emine Hafize, Assistant Professor, Kecioren Education and Training Hospital
Organization: Kecioren Education and Training Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: B.10.4.İSM.4.06.68.49/
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Alkaline Phosphatase Deficiency; Vitamin D Deficiency
Keywords: Alkaline phosphatase; Vitamin D Deficiency
MeSH Terms: conditions — Hypophosphatasia; Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Prospective study.
Masking Description: not able
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum Alp Levels In Healthy Turkish Children (Other): This study has been proceeded on children, who have no history for a chronic diseasse or medication and attending to the Keçiören Education and Research Hospital Pediatric Policlinic for routine control between September 2012-September 2013
  Interventions: Other: Serum Alkaline Phosphatase Levels

INTERVENTIONS:
Other: Serum Alkaline Phosphatase Levels — Venous blood was drawn from the patients

SUMMARY:
Alkaline phosphatase (ALP), is a metalloenzyme of the plasma membrane. Serum ALP levels in children are closely related to age and gender, many commercial test kits being used in hospitals, are only offering reference values for adults. The aim of this study is to determine serum ALP levels regarding to age, gender and pubertal stage.

DETAILED DESCRIPTION:
Alkaline phosphatase (ALP), is a metalloenzyme of the plasma membrane. Serum ALP levels in children are closely related to age and gender, many commercial test kits being used in hospitals, are only offering reference values for adults. The aim of this study is to determine serum ALP levels regarding to age, gender and pubertal stage Methods: This stuy has been proceeded on children, who have no history for a chronic diseasse or medication and attending to the Keçiören Education and Research Hospital Pediatric Policlinic for routine control between September 2012-September 2013. In order to determine the serum Alkaline Phosphatase levels in children, 1063 (511 male, 552 female) patients were incorporated. Ca, P and vitamin D levels were also evaluated. The ranges of serum ALP levels in both genders according to age has been determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* Without chronic diseases

Exclusion Criteria:

* With chronic diseases

Ages: 14 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Serum Alp Levels In Healthy Turkish Children | 1 year
  mean ALP level was determined for each age and sex and minimum and maximum levels were established.

SECONDARY OUTCOMES:
Vitamin D insufficiency | 1 year
  Regarding their child hood stage, vitamin D insufficiency were established.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abhangi KK, Choudhari SR, Butala PB, Goyal SR, Yadav TG. Salivary Total Protein and Alkaline Phosphatase Activity as Biomarkers for Skeletal Maturity and Growth Prediction in Healthy Children: An In Vivo Study. Int J Clin Pediatr Dent. 2023 Jul-Aug;16(4):603-607. doi: 10.5005/jp-journals-10005-2629. PMID 37731811
- [Background] Lala V, Zubair M, Minter DA. Liver Function Tests. 2023 Jul 30. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482489/ PMID 29494096
- [Background] Lu KL, Xie SS, Liu E, Yu XM, Wang L, Yang ZY, Xiong Q, Luo XG, Yang W, Liao W, Zhang YP. Age-wise trends in alkaline phosphatase activity in 167,625 Chinese children aged 0-18 years. Clin Biochem. 2020 May;79:34-40. doi: 10.1016/j.clinbiochem.2020.03.001. Epub 2020 Mar 3. PMID 32142736
- [Background] Topal I, Gumus B. Can Bone-Specific Alkaline Phosphatase and Osteocalcine Levels Be Used to Determine the Age in Children? Am J Forensic Med Pathol. 2020 Sep;41(3):182-187. doi: 10.1097/PAF.0000000000000555. PMID 32796205